CLINICAL TRIAL: NCT00251927
Title: An Open, Randomized, Multicenter, Phase IIIB Study During 5 Years to Assess Long-term Efficacy and Tolerability of Esomeprazole Compared to Laparoscopic Anti-reflux Surgery in Adult Subjects With Gastroesophageal Reflux Disease - LOTUS.
Brief Title: Esomeprazole (NEXIUM) vs. Surgery
Acronym: LOTUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9612C00003; SH-NEG-0003
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Results first posted 2012-08-08 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Gastroesophageal Reflux
Keywords: Acid reflux disease; Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole; Surgical Procedures, Operative

ARMS (2):
- 1 (Active Comparator): Surgery
  Interventions: Procedure: Laparoscopic fundoplication (surgery)
- 2 (Experimental): Esomeprazole (NEXIUM) therapy
  Interventions: Drug: esomeprazole

INTERVENTIONS:
Drug: esomeprazole — 40 mg oral tablet administered daily
  Other Names: Nexium®
  Arms: 2
Procedure: Laparoscopic fundoplication (surgery) — Surgery
  Arms: 1

SUMMARY:
The study investigates the efficacy of long-term treatment of esomeprazole compared to anti-reflux surgery in the control of gastroesophageal reflux disease by assessing time to treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects considered suitable for surgical treatment and long-term management of esomeprazole.
* History of chronic reflux esophagitis or symptomatic GERD

Exclusion Criteria:

* History of esophageal, gastric, or duodenal surgery predicted to influence negatively on subsequent treatment within the study.
* Contraindication to the study drug.
* Pregnancy, lactating or of child-bearing potential.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2001-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Nexium Medical Sciences Director, MD, Study Director — AstraZeneca; Lars Lundell, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (59):
- Austria (3):
  - Research Site, Linz
  - Research Site, Vienna
  - Research Site, Zell am See
- Belgium (8):
  - Research Site, Brussels
  - Research Site, Brussels (Anderlecht)
  - Research Site, Brussels (Woluwé-St-Lambert)
  - Research Site, Ghent
  - Research Site, Haine-Saint-Paul
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Rimavska Sobota
- Denmark (8):
  - Research Site, Århus C
  - Research Site, Glostrup Municipality
  - Research Site, Herning
  - Research Site, Hillerød
  - Research Site, Hvidovre
  - Research Site, Kolding
  - Research Site, Odense C
  - Research Site, Viborg
- Finland (2):
  - Research Site, Kuopio
  - Research Site, Tampere
- France (7):
  - Research Site, Bordeaux
  - Research Site, Créteil
  - Research Site, Grenoble
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Nîmes
  - Research Site, Rouen
- Germany (10):
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Herne
  - Research Site, München
  - Research Site, Tübingen
  - Research Site, Wiesbaden
  - Research Site, Würzburg
- Research Site, Reykjavik, Iceland
- Italy (10):
  - Research Site, Brescia
  - Research Site, Florence
  - Research Site, Modena
  - Research Site, Monfalcone
  - Research Site, Padua
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Rozzano
  - Research Site, San Donato Milanese
  - Research Site, Torino
- Research Site, Utrecht, Netherlands
- Norway (6):
  - Research Site, Bergen
  - Research Site, Bodø
  - Research Site, Kristiansand
  - Research Site, Oslo
  - Research Site, Tromsø
  - Research Site, Trondheim
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Lund
- Research Site, Salford, United Kingdom

REFERENCES:
- [Derived] Hatlebakk JG, Zerbib F, Bruley des Varannes S, Attwood SE, Ell C, Fiocca R, Galmiche JP, Eklund S, Langstrom G, Lind T, Lundell LR; LOTUS Study Group. Gastroesophageal Acid Reflux Control 5 Years After Antireflux Surgery, Compared With Long-term Esomeprazole Therapy. Clin Gastroenterol Hepatol. 2016 May;14(5):678-85.e3. doi: 10.1016/j.cgh.2015.07.025. Epub 2015 Jul 27. PMID 26226096
- [Derived] Attwood SE, Ell C, Galmiche JP, Fiocca R, Hatlebakk JG, Hasselgren B, Langstrom G, Jahreskog M, Eklund S, Lind T, Lundell L. Long-term safety of proton pump inhibitor therapy assessed under controlled, randomised clinical trial conditions: data from the SOPRAN and LOTUS studies. Aliment Pharmacol Ther. 2015 Jun;41(11):1162-74. doi: 10.1111/apt.13194. Epub 2015 Apr 10. PMID 25858519
- [Derived] Lundell L, Hatlebakk J, Galmiche JP, Attwood SE, Ell C, Fiocca R, Persson T, Nagy P, Eklund S, Lind T. Long-term effect on symptoms and quality of life of maintenance therapy with esomeprazole 20 mg daily: a post hoc analysis of the LOTUS trial. Curr Med Res Opin. 2015 Jan;31(1):65-73. doi: 10.1185/03007995.2014.980500. Epub 2014 Oct 31. PMID 25350223
- [Derived] Fiocca R, Mastracci L, Attwood SE, Ell C, Galmiche JP, Hatlebakk J, Barthel A, Langstrom G, Lind T, Lundell L; LOTUS trial collaborators. Gastric exocrine and endocrine cell morphology under prolonged acid inhibition therapy: results of a 5-year follow-up in the LOTUS trial. Aliment Pharmacol Ther. 2012 Nov;36(10):959-71. doi: 10.1111/apt.12052. Epub 2012 Sep 23. PMID 22998687
- [Derived] Galmiche JP, Hatlebakk J, Attwood S, Ell C, Fiocca R, Eklund S, Langstrom G, Lind T, Lundell L; LOTUS Trial Collaborators. Laparoscopic antireflux surgery vs esomeprazole treatment for chronic GERD: the LOTUS randomized clinical trial. JAMA. 2011 May 18;305(19):1969-77. doi: 10.1001/jama.2011.626. PMID 21586712

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on 16 October 2001. Last patient completed the last visit on 07 April 2009.
Pre-assignment Details: The study started with a 12-week run-in period. Patients had either been treated or untreated with a proton pump inhibitor (PPI) prior to entering this phase of the study.
Groups:
- Esomeprazole Surgical Arm: Esomeprazole 40 mg once daily during a 12-week run-in period, followed by laparoscopic anti-reflux fundoplication anti-reflux surgery.
- Esomeprazole Medical Arm: Esomeprazole 40 mg once daily during a 12-week run-in period, followed by esomeprazole treatment (start dose 20 mg once daily, if needed adjusted to 40 mg once daily)
Period: Overall Study
Arm/Group | Esomeprazole Surgical Arm | Esomeprazole Medical Arm
Started | 288 (Randomised) | 266 (Randomised)
Completed | 180 (Completed 5 year visit) | 192 (Completed 5 year visit)
Not Completed | 108 | 74
Not completed — Adverse Event | 3 | 15
Not completed — Lack of Efficacy | 22 | 16
Not completed — Lost to Follow-up | 22 | 8
Not completed — Protocol Violation | 1 | 2
Not completed — Pregnancy | 2 | 0
Not completed — Withdrawal by Subject | 40 | 25
Not completed — Study-specific discont. achieved | 13 | 2
Not completed — Study procedure non-compliance | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole Surgical Arm | Esomeprazole Medical Arm | Total
Number analyzed (Participants) | 288 | 266 | 554
Age Continuous [Mean (Standard Deviation); unit: Years] | 44.8 (10.9) | 45.3 (11.5) | 45.05 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 67 | 156
  Male | 199 | 199 | 398

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Failure at 5 Years
Description: Treatment failure in the surgical arm defined when need for medical treatment for control of symptoms from reflux disease. Treatment failure in the medical arm defined when need for treatment other than esomeprazole for control of symptoms of reflux disease.
Time Frame: During 5 years
Measure: Number; unit: participants
Arm/Group | Esomeprazole Surgical Arm | Esomeprazole Medical Arm
Number analyzed (Participants) | 288 | 266
participants | 33 | 19

2. Secondary Outcome: Los Angeles (LA) Grade 'Normal' at 5 Year Visit
Description: Endoscopic findings classified according to the Los Angeles classification:
  Grade Normal - endoscopy reveals no mucosal break Grade A- one or more mucosal breaks <5 mm in maximal length Grade B - one or more mucosal breaks >5 mm, but without continuity across mucosal folds Grade C - Mucosal breaks continuous between >2 mucosal folds, but involving less than 75% of the esophageal circumference Grade D - Mucosal breaks involving more than 75% of the esophageal circumference
Time Frame: At 5 year visit
Measure: Number; unit: participants
Arm/Group | Esomeprazole Surgical Arm | Esomeprazole Medical Arm
Number analyzed (Participants) | 288 | 266
participants | 144 | 158

3. Secondary Outcome: Investigator-assessed Heartburn Severity at 5 Year Visit, Participants With no Heartburn
Description: Presence of heartburn assessed retrospectively by the investigator. Classified by severity (none, mild, moderate, severe) Participants with no heartburn
Time Frame: At 5 year visit
Measure: Number; unit: participants
Arm/Group | Esomeprazole Surgical Arm | Esomeprazole Medical Arm
Number analyzed (Participants) | 288 | 266
participants | 163 | 161

4. Secondary Outcome: Total Score for Microscopic Reflux-related Changes in the Distal Esophagus 2 cm Above the Z-line, at 5 Year Visit
Description: The total score expressed as a mean of all the scores/number of lesions assessed; scored 2 when erosion/necrosis is found. The score could range from 0 to 2 (maximum severity). Only participants with biopsy at 5 years visit included
Time Frame: At 5 year visit
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Esomeprazole Surgical Arm | Esomeprazole Medical Arm
Number analyzed (Participants) | 153 | 177
units on a scale | 0.23 (0.10) | 0.25 (0.03)

5. Secondary Outcome: Percentage Time With pH<4 During 24-hour pH Metry at 5 Year Visit
Description: Intra-gastric acid exposures assessed by 24-h pH-metry. Only participants with pH-emtry performed at 5 year visit included
Time Frame: At 5 year visit
Measure: Mean (Standard Deviation); unit: percentage of time recorded
Arm/Group | Esomeprazole Surgical Arm | Esomeprazole Medical Arm
Number analyzed (Participants) | 124 | 162
percentage of time recorded | 2.9 (7.0) | 4.7 (7.0)

6. Secondary Outcome: Los Angeles (LA) Grade 'A' at 5 Year Visit
Description: as for outcome 2
Time Frame: At 5 year visit
Measure: Number; unit: participants
Arm/Group | Esomeprazole Surgical Arm | Esomeprazole Medical Arm
Number analyzed (Participants) | 288 | 266
participants | 12 | 16

7. Secondary Outcome: Los Angeles (LA) Grade 'B' at 5 Year Visit
Description: as for outcome 2
Time Frame: At 5 year visit
Measure: Number; unit: participants
Arm/Group | Esomeprazole Surgical Arm | Esomeprazole Medical Arm
Number analyzed (Participants) | 288 | 266
participants | 5 | 7

8. Secondary Outcome: Los Angeles (LA) Grade C at 5 Year Visit
Description: as for outcome 2
Time Frame: At 5 year visit
Measure: Number; unit: participants
Arm/Group | Esomeprazole Surgical Arm | Esomeprazole Medical Arm
Number analyzed (Participants) | 288 | 266
participants | 1 | 2

9. Secondary Outcome: Investigator-assessed Heartburn Severity at 5 Year Visit, Participants With Mild Heartburn
Description: Presence of heartburn assessed retrospectively by the investigator. Classified by severity (none, mild, moderate, severe). Participants with mild heartburn
Time Frame: At 5 year visit
Measure: Number; unit: participants
Arm/Group | Esomeprazole Surgical Arm | Esomeprazole Medical Arm
Number analyzed (Participants) | 288 | 266
participants | 11 | 25

10. Secondary Outcome: Investigator-assessed Heartburn Severity at 5 Year Visit, Participants With Moderate Heartburn
Description: Presence of heartburn assessed retrospectively by the investigator. Classified by severity (none, mild, moderate, severe). Participants with moderate heartburn
Time Frame: At 5 year visit
Measure: Number; unit: participants
Arm/Group | Esomeprazole Surgical Arm | Esomeprazole Medical Arm
Number analyzed (Participants) | 288 | 266
participants | 3 | 3

11. Secondary Outcome: Investigator-assessed Heartburn Severity at 5 Year Visit, Participants With Severe Heartburn
Description: Presence of heartburn assessed retrospectively by the investigator. Classified by severity (none, mild, moderate, severe). Participants with severe heartburn
Time Frame: At 5 year visit
Measure: Number; unit: participants
Arm/Group | Esomeprazole Surgical Arm | Esomeprazole Medical Arm
Number analyzed (Participants) | 288 | 266
participants | 0 | 2

ADVERSE EVENTS:
Groups:
- Non-Surgical Arm: This group of patients was randomized to receive surgery but were on operated on and were followed for safety purposes
Arm/Group | Esomeprazole Surgical Arm | Esomeprazole Medical Arm | Non-Surgical Arm
Serious Adverse Events (participants affected / at risk) | 103/248 | 101/266 | 3/40
Other Adverse Events (participants affected / at risk) | 0/248 | 0/266 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole Surgical Arm (N=248) | Esomeprazole Medical Arm (N=266) | Non-Surgical Arm (N=40)
Microcytic Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 2 | 0
Angina Pectoris (Cardiac disorders) | 1 | 3 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 1
Cardiac Failure (Cardiac disorders) | 0 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 2 | 0 | 0
Coronary Artery Stenosis (Cardiac disorders) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 3 | 0
Myocardial Ischaemia (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0 | 0
Conductive Deafness (Ear and labyrinth disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Corneal Oedema (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Keratitis (Eye disorders) | 0 | 1 | 0
Retinal Vein Occlusion (Eye disorders) | 1 | 0 | 0
Abdominal Hernia (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0
Acute Abdomen (Gastrointestinal disorders) | 0 | 1 | 0
Barrett's Oesophagus (Gastrointestinal disorders) | 1 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Colonic Pseudo-Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diverticulitis Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gastric Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Gastric Ulcer Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis Haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Ileus Paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 | 0 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 1 | 0
Lumbar Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0
Chest Discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Dysplasia (General disorders) | 1 | 0 | 0
Multi-Organ Failure (General disorders) | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 3 | 5 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Bile Duct Stenosis (Hepatobiliary disorders) | 0 | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 2 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 0 | 0
Abscess Jaw (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 2 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 3 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0
Pneumonia Primary Atypical (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Tubo-Ovarian Abscess (Infections and infestations) | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 0
Complication Of Device Insertion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gas Poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 3 | 0 | 0
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Operative Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 4 | 0 | 0
Procedural Complication (Injury, poisoning and procedural complications) | 2 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 3 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skull Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0
Urinary Bladder Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 2 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign Neoplasm Of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign Peritoneal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carcinoid Tumour Pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant Neoplasm Of Spermatic Cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tongue Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 1 | 0 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 2 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0 | 0
Anxiety Disorder (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 0
Calculus Ureteric (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 2 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian Torsion (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine Polyp (Reproductive system and breast disorders) | 1 | 1 | 0
Vaginal Prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Suffocation Feeling (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vocal Cord Cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Skin Fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 2 | 0
Arterial Thrombosis Limb (Vascular disorders) | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 1 | 0
Necrosis Ischaemic (Vascular disorders) | 0 | 1 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 1 | 0
Varicose Vein (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No